CLINICAL TRIAL: NCT03868748
Title: Safety Evaluation of β-arbutin in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SP Nutraceuticals Inc. (Industry)
Collaborators: Canadian Glycomics Network (GlycoNet) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 241603
Record Dates: First submitted 2018-11-20; First posted 2019-03-11 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Arbutin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): The double-blind phase of the study starts with randomized allocation of eligible participants to one of three treatment arms. Participants randomized to the placebo treatment arm will consume one placebo capsule per day for 12 weeks
  Interventions: Other: Placebo
- Low Dose, 12 weeks (Experimental): The double-blind phase of the study starts with randomized allocation of eligible participants to one of three treatment arms. Participants randomized to the low dose treatment arm will consume one 150 mg beta-arbutin capsule per day for 12 weeks.
  Interventions: Dietary Supplement: Beta-arbutin; Other: Placebo
- High Dose, 4 weeks (Experimental): The double-blind phase of the study starts with randomized allocation of eligible participants to one of three treatment arms. Participants randomized to the high dose treatment arm will consume one placebo capsule per day for 8 weeks followed by one 400 mg beta-arbutin capsule per day for 4 weeks.
  Interventions: Dietary Supplement: Beta-arbutin; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-arbutin — Beta-arbutin capsules
  Other Names: SP001
  Arms: High Dose, 4 weeks; Low Dose, 12 weeks
Other: Placebo — Placebo capsules containing non-medicinal ingredients

SUMMARY:
The purpose of this study is to determine the safety of synthetic beta-arbutin, a dietary supplement that aids in the prevention and treatment of calcium oxalate kidney stones, when administered to healthy human subjects.

DETAILED DESCRIPTION:
The objective and purpose of this Phase I study is to investigate the safety of synthetic beta-arbutin, administered to healthy human subjects for: i) 12 weeks, at a dose of 150 mg/day, and ii) 4 weeks, at a dose of 400mg/day. Safety will be determined by assessing adverse event rates between treatment groups and mean changes relative to baseline in serum biochemical, hematological and urinary markers.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 18-65 years
* includes non-pregnant, non-breastfeeding women on adequate birth control
* acceptable effective contraceptive methods for participants with child-bearing potential include: barrier methods (condoms), total abstinence, hormonal birth control methods (oral, injectable, transdermal, or intra-vaginal), intrauterine devices, and confirmed successful vasectomy of partner;
* Body Mass Index (BMI) of 18.5-35 kg/m2;
* Generally healthy (absence of active clinical disease as determined by serum biochemical, hematological, and urinary parameter tests as well as detailed medical history and blood pressure measurements) as assessed by the PI/QI;
* Males and females of childbearing potential willing to use appropriate effective contraception for the duration of the study;
* Agrees to maintain current diet and exercise routine during the study;
* Ability to provide written informed consent; and
* Willing to comply with all study requirements and provide urine and blood specimens over the 12-week study period..

Exclusion Criteria:

* Pregnant or breastfeeding women;
* History of renal dysfunction;
* History of macular degeneration as assessed by the PI/QI;
* History of liver disease as assessed by the PI/QI;
* Type I or Type II diabetes;
* Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the PI/QI History of renal dysfunction, as assessed by the PI/QI;
* Cancer being actively treated with systemic therapy (i.e. chemotherapy, immune therapy);
* Self-reported HIV-, Hepatitis B-, and/or C-positive diagnosis;
* High alcohol intake (average of > 2 standard drinks per day);
* Heavy smokers (average of >10 cigarettes per day);
* Use of cannabinoid products within 30 days of enrollment;
* Any history of major surgery (i.e. inter-abdominal, inter-thoracic, inter-cranial) within the last six months, or surgery planned during the course of the study;
* Known hypersensitivity to arbutin;
* Allergy to all ingredients (including non-medicinal ingredients) in investigational products and placebo product
* Self-reported medical or neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation; and
* Clinically significant abnormal laboratory results at screening as assessed by the PI/QI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AE) | During treatment period (Day 1 to Day 84)
  Number of treatment emergent adverse events according to CTCAE v5.0.

SECONDARY OUTCOMES:
Participant compliance to treatment | During treatment period (day 7, day 28, day 56, day 84)
  Adherence to study protocol and study product consumption as ascertained by capsule counts
Hematology | At screening and during treatment period (day 7, day 28, day 56, day 84)
  Number of clinically relevant changes in hematology markers as assessed by: hematocrit (HCT), hemoglobin (Hb), red blood cell count (RBC), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), white blood cell count (WBC), differential blood count (neutrophils, lymphocytes, monocytes, eosinophils and basophils), reticulocytes absolute count, and mean platelet volume (MPV). Assessments will be performed at screening and during treatment period.
Biochemistry | At screening and during treatment period (day 7, day 28, day 56, day 84)
  Number of clinically relevant changes in serum biochemistry. Enzymes: aspartate transaminase, alanine transaminase, alkaline phosphatase, gamma amyl transferase. Electrolytes: magnesium, sodium, potassium, chloride, calcium. Substrates: glucose (non-fasted), bilirubin (total, direct and indirect), creatinine, albumin, urea, vitamin D. Hormones: parathyroid hormone, thyroid stimulating hormone (TSH). Coagulation tests: international normalized ratio (INR), partial thromboplastin time (PTT). Assessments will be performed at screening and during treatment period.
Urinalysis (Routine) | At screening and during treatment period (day 7, day 28, day 56, day 84)
  Number of clinically relevant changes in routine dipstick urinalysis which will assess: pH, specific gravity, protein, glucose, ketones, blood, nitrite, and bilirubin. Assessments will be performed at screening and during treatment period.
Urinalysis (Microscopy) | At screening and during treatment period (day 7, day 28, day 56, day 84)
  Microscopy (RBC, WBC and casts [Hyaline, Granular and Cellular]) by thermodilatometry (TDL) may be performed at additional urinalysis time points if clinically relevant abnormalities are detected (positive result for protein or blood in dipstick). Assessments will be performed at screening and during treatment period.
Urine culture | At screening and during treatment period (day 7, day 28, day 56, day 84)
  Urine culture will be performed to detect microorganisms. Assessments will be performed at screening and during treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Razvi, MD, FRCSC, Principal Investigator — Chair/Chief, Division of Urology; David Crowley, MD, Principal Investigator — KGK Science site qualified investigator
Locations (2):
- Canada (2):
  - St Joseph's Health Care London, St. Joseph's Hospital, London, Ontario
  - KGK Science, London, Ontario

IPD SHARING:
Plan to Share IPD: No